CLINICAL TRIAL: NCT00316797
Title: Phase 1 Assessment of the Biodistribution and Safety of 123-I INER in Healthy Subjects
Brief Title: Biodistribution and Safety of a Radiopharmaceutical in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: Molecular NeuroImaging (Other)
Responsible Party: Principal Investigator, John Seibyl, MD, Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: H01_INER_001/002
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Neurodegenerative Diseases
Keywords: SPECT; Nuclear Medicine
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 123-I INER (Experimental): To assess 123-I INER
  Interventions: Drug: 123-I INER

INTERVENTIONS:
Drug: 123-I INER — Serial whole body planar imaging in the anterior and posterior projection will be performed at 1 min, 30 min, 1 h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, and 18-24h following injection of 5 mCi of 123-I INER. Venous blood data will be acquired at each imaging time point. In addition a 24 hour urine collection will commence following radiotracer injection and urine sampled in five collections every 4 hours collection for first sixteen hours (4 collections), then one collection from 16 to 24 h. Whole body and source organs uptake will be analyzed on anterior and posterior images for calculating the radiation absorbed doses to organs using the MIRD method as described previously (Seibyl, et al, 1993). Plasma and urine metabolites will be characterized and safety assessments obtained.

SUMMARY:
The initial study of [123I] INER will be completed in two parts. Once Part A (Preliminary whole body biodistribution) is completed, Part B (Serial dynamic SPECT assessment of regional brain uptake and washout and plasma metabolite analysis to determine the brain penetrance and regional distribution and washout counts following 123-I INER injection) will commence. All study procedures will be conducted at the Institute for Neurodegenerative Disorders (IND) and Molecular NeuroImaging (MNI) in New Haven, CT. All subjects will undergo written informed consent and a screening evaluation including baseline clinical laboratory testing, and a baseline physical and neurological evaluation.

DETAILED DESCRIPTION:
All subjects will receive a full physical examination at IND to determine study eligibility. Written informed consent will be obtained prior to any study procedures. The screening procedures will include: review of medical and psychiatric history, review of medications, physical examination including height and body weight, vital sign measurements, review of inclusion/exclusion criteria, clinical laboratory testing (serum chemistries, CBC, urinalysis, urinary drug screen), urine pregnancy test for females of childbearing potential and electrocardiogram in preparation for the imaging study.

Part A: Four healthy subjects will each receive one injection of 123-I INER. Serial whole body planar imaging in the anterior and posterior projection will be performed over the 8-9 hour period following injection of 5 mCi of 123-I INER and again at 18-24 hours following injection. Venous blood data will be acquired at each imaging time point. In addition a 24 hour urine collection will commence following radiotracer injection. Whole body and source organs uptake will be analyzed on anterior and posterior images for calculating the radiation absorbed doses to organs. Plasma and urine metabolites will be characterized and safety assessments obtained. Serial safety assessments will include vital signs, serum chemistries, CBC, urinalysis, and EKGs.

Part B: Six healthy subjects will each receive one injection of 123-I INER. Following bolus intravenous injection of 5 mCi of 123-I INER over 15 seconds, serial dynamic SPECT brain acquisitions will be obtained to evaluate the regional brain uptake and washout of activity. Venous blood measures will be obtained with each acquisition and characterization of 123-I INER and metabolites will be assessed. Safety assessments will include vital signs, serum chemistries, CBC, urinalysis, and EKGs.

ELIGIBILITY:
Inclusion Criteria:

* The subject is aged 18-65.
* Written informed consent is obtained.
* The subject has a negative history of neurological or psychiatric illness based on evaluation by a research physician.
* For females, non-child bearing potential or negative urine pregnancy test on day of [123I] INER injection.

Exclusion Criteria:

* The subject has a clinically significant clinical laboratory values abnormality, and/or medical or psychiatric illness.
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery).
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Use of all prescription drugs or non-prescriptions drugs that may effect norepinephrine such as cold remedies (for 2 weeks prior to injection).
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-04; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Assess the biodistribution and metabolic rate of 123-I INER for determination of radiation absorbed dose estimates. | 2 yrs

SECONDARY OUTCOMES:
Assess of regional brain uptake and washout and plasma metabolite analysis to determine the brain penetrance and regional distribution and washout counts following 123-I INER injection. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John Seibyl, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

REFERENCES:
- [Background] Abi-Dargham A, Innis RB, Wisniewski G, Baldwin RM, Neumeyer JL, Seibyl JP. Human biodistribution and dosimetry of iodine-123-fluoroalkyl analogs of beta-CIT. Eur J Nucl Med. 1997 Nov;24(11):1422-5. doi: 10.1007/s002590050170. PMID 9371877
- [Background] Dey HM, Seibyl JP, Stubbs JB, Zoghbi SS, Baldwin RM, Smith EO, Zubal IG, Zea-Ponce Y, Olson C, Charney DS, et al. Human biodistribution and dosimetry of the SPECT benzodiazepine receptor radioligand iodine-123-iomazenil. J Nucl Med. 1994 Mar;35(3):399-404. PMID 8113883
- [Background] Fujita M, Seibyl JP, Vaupel DB, Tamagnan G, Early M, Zoghbi SS, Baldwin RM, Horti AG, KoreN AO, Mukhin AG, Khan S, Bozkurt A, Kimes AS, London ED, Innis RB. Whole-body biodistribution, radiation absorbed dose, and brain SPET imaging with [123i]5-i-A-85380 in healthy human subjects. Eur J Nucl Med Mol Imaging. 2002 Feb;29(2):183-90. doi: 10.1007/s00259-001-0695-z. PMID 11926380
- [Background] Seibyl JP, Wallace E, Smith EO, Stabin M, Baldwin RM, Zoghbi S, Zea-Ponce Y, Gao Y, Zhang WY, Neumeyer JL, et al. Whole-body biodistribution, radiation absorbed dose and brain SPECT imaging with iodine-123-beta-CIT in healthy human subjects. J Nucl Med. 1994 May;35(5):764-70. PMID 8176456
- See also: Institute for Neurodegenerative Disorders — http://www.indd.org